CLINICAL TRIAL: NCT05711368
Title: The Effects of Distress Tolerance Training on Problematic Internet Use and Psychological Wellbeing Among Faculty Nursing Students
Brief Title: Effect of Distress Tolerance Training on Problematic Internet Use and Psychological Wellbeing Among Faculty Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, ayman el-ashry, lecturer at psychiatric and mental health nursing, faculty of nursing, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00013620/9/2022/48
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Nurse's Role
Keywords: Distress Tolerance; Problematic Internet Use; Psychological well being; Nursing
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Active Comparator): Nursing students who participated in distress tolerance training session
  Interventions: Behavioral: Distress tolerance training
- control group (No Intervention): Nursing students not participating in distress tolerance training session

INTERVENTIONS:
Behavioral: Distress tolerance training — It consisted of seven sessions. A 90-minute session will be conducted twice a week for four weeks. The first introductory session will be concerned with helping the student learn how to engage in distress tolerance training and define goals of distress tolerance. At the end of the 1st session, a written plan for every session (time, duration and setting) will be scheduled individually with each student.The next six training sessions will cover three core skills which comprised three sets: Crisis Survival Skills, the skills of Reality Acceptance; and the Skills When the Crisis Is Addiction. The distress tolerance training methods will include individualized interactions, demonstration, and rehearsal, psychoeducation, practice exercises and homework assignments. Follow up between sessions will done using telephone calling and messaging in order to encourage performance homework assignments, and provide help and support when needed particularly at the time of stress. .
  Other Names: dialectical behavioral therapy
  Arms: interventional group

SUMMARY:
The Internet is a social environment as well as a tool. In this digital environment, where students interact with each other, live, and generally comprehend their cultures, college students learn information. The Internet has become essential to college students' daily lives and education. The World Health Organization (WHO) has cautioned that increased screen usage and gaming may occur during the COVID-19 pandemic. Due to this, there is an increased chance of Internet and gaming addiction, leading to more distress and concern for students' psychological well-being. Therefore, university students needed an intervention program to overcome these problems. The researchers in the present study will use distress tolerance. Distress tolerance (DT) is defined as one's ability to continue engaging in goal-directed behavior in the face of emotional, cognitive, or physical discomfort. Eventually, the present study aimed to The present study aims to:

Assess the impact of distress tolerance training on problematic internet use and psychological wellbeing among university nursing students.

Research Hypothesis:

Nursing students who receive distress tolerance training will exhibit lower problematic internet use and better psychological wellbeing than those who didn't receive it

ELIGIBILITY:
Inclusion Criteria:

* Students that are not participating in any other type of psychotherapy.
* Students who scored high on Problematic Internet Use Questionnaire (PIU).

Exclusion Criteria:

* Students who have a history of mental illness.
* students who are more than 30 years old.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
The Problematic Internet Use Questionnaire (PIU) | up to 16 weeks
  The Problematic Internet Use Questionnaire was developed by and it is an 18-item self- report scale that measures the extent of how risky internet usage can be. Items are scored from 1 = never to 5 = always. This test has three factors, i.e., Obsession, Neglect, and Control disorder. Earlier studies showed that PIU subscales have good psychometric properties, with high reliability (αs of .74-.87), high 3-week stability (rs from .76 to .90), and acceptable discriminant validity (e.g., confirmed by negligible associations with alcohol or illicit drug use and significant but weak associations with the use of gaming machines).
Ryff psychological well being scale (PWBS) | up to 16 weeks
  The Ryff psychological well being scale was originally consisted of six 7-item subscales for the assessment of six factors: (1) autonomy; (2) environmental mastery; (3) personal growth; (4) positive relations with others; (5) purpose in life and (6) self-acceptance. Response categories for these items are scored along a seven-point Likert scale ranging from strongly disagree (1) to strongly agree (7). The scores of some items will be reversed as recommended in Ryff's original PWBS. The scores for six subscales were calculated as averages; higher mean scores indicate greater psychological wellbeing. Internal consistency (alpha coefficients) was estimated from a sample of older and middle-aged groups , average alphas were .78, and .77, respectively, for the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demetrovics Z, Szeredi B, Rozsa S. The three-factor model of Internet addiction: the development of the Problematic Internet Use Questionnaire. Behav Res Methods. 2008 May;40(2):563-74. doi: 10.3758/brm.40.2.563. PMID 18522068
- [Background] Gao J, McLellan R. Using Ryff's scales of psychological well-being in adolescents in mainland China. BMC Psychol. 2018 Apr 20;6(1):17. doi: 10.1186/s40359-018-0231-6. PMID 29678202
- [Background] Leyro TM, Zvolensky MJ, Bernstein A. Distress tolerance and psychopathological symptoms and disorders: a review of the empirical literature among adults. Psychol Bull. 2010 Jul;136(4):576-600. doi: 10.1037/a0019712. PMID 20565169
- [Background] Gong Z, Wang L, Wang H. Perceived Stress and Internet Addiction Among Chinese College Students: Mediating Effect of Procrastination and Moderating Effect of Flow. Front Psychol. 2021 Jun 28;12:632461. doi: 10.3389/fpsyg.2021.632461. eCollection 2021. PMID 34262501